CLINICAL TRIAL: NCT03546101
Title: Early Detection of Epstein-Barr Virus Related Disease. Improving Quantification of EBV in Blood Samples Using Polymerase Chain Reaction.
Brief Title: Early Detection of Epstein-Barr Virus Related Disease.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EBV-KMA; 1-16-02-685-16 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2018-05-07; First posted 2018-06-06 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-12

CONDITIONS: Post-transplant Lymphoproliferative Disorder; Mononucleosis; Epstein-Barr Virus Infections; Epstein-Barr Virus Related Malignancy; Epstein-Barr Viraemia; Epstein-Barr Virus-Related Hodgkin Lymphoma; Epstein-Barr Virus-Related Non-Hodgkin Lymphoma; Hemophagocytic Lymphohistiocytoses; Hemophagocytosis
MeSH Terms: conditions — Infectious Mononucleosis; Epstein-Barr Virus Infections; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Department of Kidney Medicine: Primarily transplant recipients undergoing monitoring for EBV and patients suspected for having PTLD.
- Department of Hematology: Patients diagnosed with PTLD and other kinds of lymphoma. Patients undergoing hematopoietic stem cell transplantation and patients with hemophagocytosis.
- Department of pediatrics: Children undergoing transplantation. Children diagnosed with hemophagocytic lymphohistiocytosis.

SUMMARY:
Epstein-Barr virus (EBV) is one of several herpesviruses that cause disease in humans. EBV virus has an oncogenic potential, and it has been associated with the development of a wide range of cancers. Previous studies have shown a close association between EBV and Post-Transplant Lymphoproliferative disorder (PTLD) in transplant recipients. As part of a preventive approach against PTLD, several transplantation units now monitor the occurrence of EBV-DNAemia after transplantation. However, there is little evidence to guide this strategy; nor is there consensus concerning either the best specimen to use for EBV analysis (whole blood or plasma).

In this study investigators aim to optimise and validate a polymerase chain reaction (PCR)-test for EBV-DNA on, respectively, whole blood, plasma and a combination of plasma and lymphocytes.

The investigators wish to determine which of the three tests best predicts current and future risk of development of EBV-related diseases such as mononucleosis and PTLD.

DETAILED DESCRIPTION:
EBV is one of several herpesviruses that cause disease in humans. Primary EBV infection usually occurs in early childhood and is generally asymptomatic, while later infection may cause mononucleosis. As with other herpesviruses, primary infection is followed by persistent (lifelong) infection. EBV virus has an oncogenic potential, and it has been associated with the development of a wide range of cancers. Previous studies have shown a close association between EBV and PTLD in transplant recipients. As part of a preventive approach against PTLD, several transplantation units now monitor the occurrence of EBV-DNAemia after transplantation. However, there is little evidence to guide this strategy; nor is there consensus concerning either the best specimen to use for EBV analysis (whole blood or plasma) or the appropriate clinical action to take if EBV-DNAemia is detected.

In this study investigators aim to optimise and validate a polymerase chain reaction (PCR)-test for EBV-DNA on, respectively, whole blood and a combination of plasma and lymphocytes.

Results obtained with the two new methods will be compared with those from the already established World Health Organization (WHO) standardised EBV-PCR test on ethylenediaminetetraacetic acid (EDTA)-plasma. The result of all three tests will be evaluated relative to EBV-related symptoms and other diseases.

The investigators wish to determine which of the three tests best predicts current and future risk of development of EBV-related diseases such as mononucleosis and PTLD.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected for having EBV disease.

Exclusion Criteria:

* If the patients has any contraindications for blood sampling.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Transplant recipients undergoing monitoring for EBV and patients suspected or diagnosed with PTLD.
  Patients undergoing hematopoietic stem cell transplantation and patients with hemophagocytosis.
  Children undergoing transplantation. Children diagnosed with hemophagocytic lymphohistiocytosis.
Sampling Method: Non-Probability Sample
Enrollment: 1527 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of proven EBV disease | From time of blood sampling up to 24 months.
  Symptoms compatible with EBV disease combined with a tissue biopsy positive for EBV
Incidence of probable EBV disease | From time of blood sampling up to 24 months.
  Symptoms compatible with EBV disease combined with a positive EBV-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Lene Ugilt, MD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Central Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ludvigsen LUP, Andersen AS, Hamilton-Dutoit S, Jensen-Fangel S, Bottger P, Handberg KJ, Ivarsen P, d'Amore F, Bibby BM, Albertsen BK, Jespersen B, Thomsen MK. A prospective evaluation of the diagnostic potential of EBV-DNA in plasma and whole blood. J Clin Virol. 2023 Oct;167:105579. doi: 10.1016/j.jcv.2023.105579. Epub 2023 Aug 30. PMID 37683299